CLINICAL TRIAL: NCT03456050
Title: Effectiveness of a New Therapeutic Technique 'Functional Range Conditioning' in Treating Patients With Chronic Non-specific Low Back Pain
Brief Title: Effectiveness of 'Functional Range Conditioning' in Treating Patients With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Reem S. Alattallah, Post Graduate student, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAMS 028-3839
Record Dates: First submitted 2018-02-26; First posted 2018-03-07 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Outcome provider masked about the outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FRC group (Experimental): This group will receive FRC exercise.
  Interventions: Behavioral: FRC exercise
- Conventional treatment (Experimental): This group will receive conventional exercise.
  Interventions: Behavioral: Conventional Exercise

INTERVENTIONS:
Behavioral: FRC exercise — The program will consist of hip joint controlled articular rotations (CARs) in standing position for 3 - 5 repetitions. Then, the participant will sit on the floor in what is called 90/90 position which is sitting in hip and flexion in 90 degrees for both the lead (front) and trail (side) leg. The participant will perform a Progressive and regressive angular isometric loadings (PAILs and RAILs) for the trail leg to increase the range of internal rotation, the contraction will be performed three times and the holding of the position will be for two minutes. After expanding the range, the participant will perform Progressive and regressive angular loadings (PALs and RALs) isometric contractions in form of a passive range hold for internal rotation and abduction, for 3 - 5 times.
  Arms: FRC group
Behavioral: Conventional Exercise — The conventional training program in this study will be the routine training for increasing the hip rotation. By screening the scientific literature, the conventional training found to consists of static stretching and strengthening using body weight and/or a band and the time of holding a stretch is about 30 seconds. For that the flexibility exercise will consist of progressive stretching from a prone position (leg fall in a stretch), the participant will perform 3 - 5 repetitions with 30 seconds hold or as tolerated. The strengthening exercise consists of hip abduction (hip opening) using a band or ankle weight from side lying for 10 - 12 repetitions 3 times.
  Arms: Conventional treatment

SUMMARY:
The aims of this study are to examine the effectiveness of functional range conditioning in patients with chronic non-specific low back pain in terms of improving hip internal rotation and strength of the hip abductors, and reducing pain and disability.

DETAILED DESCRIPTION:
It will be a single blind two-arm randomized controlled trial. Saudi men and women aged between 25 - 45 years with a diagnosis of chronic non-specific low back pain will be invited to participate in this study. Subjects who will fulfill the study's criteria and who are willing to participate in this study will be asked to sign an informed consent form. The primary outcome will be the active and passive range of motion (ROM) of the hip internal rotators and it will be measured using digital inclinometer. The secondary outcomes in this study will be the maximum torque of the hip abductors (gluteus medius), concentric at a constant, low-speed, and high-speed. The peak torque and strength will be measured using isokinetic dynamometry, pain intensity will be assessed using a visual analog scale and disability will be assessed using Oswestry disability index. All participants will have their information taken by the principal investigator. Subsequently, participants will randomly be assigned to either the FRC group or the conventional treatment group by the principal investigator. Concealed randomization will be performed by means of a computer-generated table of random numbers. Outcomes will be measured at baseline, week 4 and week 8 for all participants in both groups by an assistant researcher.

ELIGIBILITY:
Inclusion Criteria:

* Saudi men and women aged between 25 - 45 years with a diagnosis of chronic non-specific low back pain

Exclusion Criteria:

* Hip, spine and knee pathology.
* Hip and knee replacement.
* Surgery and fracture within the last 6 months.
* Cancer.
* Pregnant women.
* Any medical condition that precluded safe participation in exercise programs such as significant cardiac, pulmonary, neurological disease or mental disorder.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Passive range of motion (Hip internal rotation) | Change from baseline passive hip internal range of motion at 8 weeks
  It will be measured using digital inclinometer

SECONDARY OUTCOMES:
Strength of the hip abductors (gluteus medius) | Change from baseline hip abductors strength at 8 weeks
  Strength of the hip abductors will be measured using hand held dynamometer or isokinetic dynamometry,
Pain Intensitiy | Change from baseline pain intensity at 8 weeks
  Pain intensity will be assessed using visual analog scale (VAS) (0 - 10 cm with 0 indicates no pain and 10 indicates the worst pain).
Functional disability | Change from baseline functional disability at 8 weeks
  Functional disability will be assessed using Oswestry disability index. Each item in the questionnaire is scored on a 0-5 scale with zero indicating the least amount of disability and the 5 indicating most severe disability.The scores for total items answered are summed, and multiplied by two to get the index (range 0 to 100). Zero indicates no disability and 100 indicates maximum possible disability.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed alghadir, PHD, Study Director — King Saud University
Locations (1):
- King Saud University, Riyāḑ, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with principal investigator (Ms. Reem S. Alattallah) and sub-investigator (Dr. Ahmad Alghadir) due to confidentiality issues